CLINICAL TRIAL: NCT03631589
Title: Treatment of Steroid-resistant Severe Acute Graft-versus-host Disease With Mesenchymal Stem Cells
Brief Title: MSC for Severe aGVHD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Jianda Hu, Director of the department of Hematology, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-SCT-01
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Steroid-resistant Severe aGVHD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSCs treated (Experimental)
  Interventions: Biological: MSCs

INTERVENTIONS:
Biological: MSCs — mesenchymal stem cells therapy

SUMMARY:
Steroid-resistant acute graft-versus-host disease (aGVHD) is one of the most severe complications in the setting of allogeneic hematopoietic stem cell transplantation (HSCT), which cannot be significant benefit from the second-line therapies.The mesenchymal stem cells (MSCs) possess extensive immunomodulatory properties and are very promising to rescue the refractory aGVHD.This study aims to assess the efficacy and safety of MSCs for the treatment of the refractory aGVHD.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged <65 years
* Patients with steroid-resistant severe aGVHD
* Cardiac: Left ventricular ejection fraction ≥ 50%
* Adequate renal and hepatic function
* Performance status: Karnofsky ≥ 70%

Exclusion Criteria:

* Pregnant or lactating females.
* Any co-morbidity precluding the administration of MSCs.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
complete and partial response rate | 1 year

SECONDARY OUTCOMES:
Adverse events that are related to treatment | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China